CLINICAL TRIAL: NCT02413619
Title: Refractive Consequences of Epiretinal Membrane Surgery
Acronym: EPIREF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Hassan Hamoudi, MD, Glostrup University Hospital, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIREF
Record Dates: First submitted 2015-03-27; First posted 2015-04-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Vitrectomy; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Start cataract (Active Comparator): Patients start having cataract surgery. After one month they undergo vitrectomy
  Interventions: Procedure: Cataract surgery
- start vitrectomy (Active Comparator): Patients start having vitrectomy. After one month they undergo cataract surgery.
  Interventions: Procedure: Vitrectomy
- combined surgery (Active Comparator): Combined cataract surgery and vitrectomy at the same time
  Interventions: Procedure: Combined surgery

INTERVENTIONS:
Procedure: Vitrectomy — Vitrectomy
  Arms: start vitrectomy
Procedure: Cataract surgery — Cataract surgery
  Arms: Start cataract
Procedure: Combined surgery — Combined vitrectomy and cataract surgery at the same time
  Arms: combined surgery

SUMMARY:
Epiretinal membrane is treated with vitrectomy and peeling. Afterwards cataract is usually developed, which requires a cataract surgery.

The aim of this study is to investigate the refractive consequences of surgery for Epiretinal membrane and cataract.

Investigators investigate the sequence of surgery in patients having surgery for Epiretinal membrane and cataract in a prospective clinically randomized intervention trial. Patients are randomized to 1) start with vitrectomy, 2) start with cataract surgery, 3) combined surgery. Investigators want to find the sequence of surgery that gives the most optimal refractive result, the most stabile intraocular lens, and the minimal loss of corneal endothelial cells.

DETAILED DESCRIPTION:
Aim: To evaluate the impact of the sequence of surgery on the Refractive Error and the Corneal Endothelial Count in phakic individuals undergoing surgery for Epiretinal membrane.

Study design: Prospective interventional randomized clinical trial. Primary outcome: Refractive error (i.e. Intraocular lens power prediction error), Corneal Endothelial Count, and postoperative macular oedema.

Secondary outcome: Changes in axial length, anterior chamber depth and keratometry; the accuracy of formulas used to calculate the power of the intraocular lens.

Study population:

Identification of participants: Individuals referred to the Macular Surgery Clinic, Surgical Retina Team, Department of Ophthalmology, Glostrup University Hospital, Copenhagen, Denmark. The individuals should be signed up for surgery because of Epiretinal membrane at the clinic.

Method:

Individuals are randomized to the possible sequences of surgery (i.e. start with cataract surgery, start with vitrectomy, or combined surgery). Based on an estimated clinical relevant refractive prediction error of 0,50 diopter and a standard deviation of 0,50 diopter, a number of 20 individuals in each of the three groups are needed to obtain a power of 80 % and a type 1 error of 5 %. Total number of individuals is thus 60.

Clinical examinations are performed preoperatively and 2 weeks after each surgery (cataract surgery, vitrectomy or combined surgery), and 3 and 12 months postoperatively. The examinations include best corrected distance visual acuity, autorefraction/keratometry (Retinomax®, Nikon, Tokyo, Japan), subjective refraction, slit-lamp examination, fundoscopy and tonometry. Biometry by IOLMaster (Carl Zeiss, Meditec AG, Germany), intraocular power calculation with the SRK/T formula. Pentacam Scheimpflug Cornea tomography (Topcon, Tokyo, Japan). Corneal Endothelial Count obtained by three images of the central region of the corneal endothelium (Topcon SP-3000P, Tokyo, Japan). Heidelberg Optical Coherence Tomography, (Heidelberg Engineering, Heidelberg, Germany).

Sequence of surgery depends on randomization. In all cases a standard phacoemulsification (scleral tunnel or clear corneal incision) with in-the-bag intraocular lens implantation. In combined surgery, the cataract surgery is performed before vitrectomy during the same session. Vitreoretinal procedures include a standard three-port 23 gauge pars plana vitrectomy, membrane peeling, and the use of dyes. Cataract surgery is performed by one of two experienced surgeons, and vitrectomy is carried out by one experienced surgeon.

Analysis: A computer database will be created as a fill-in form to record all patient data, and a masked statistical analysis of all outcome measures will be performed. Statistical analysis will be performed to determine differences in baseline data among the three groups (age, sex, visual acuity, keratometry, axial length, anterior chamber depth, Corneal Endothelial Count). To identify independent predictors for all outcome measures at different follow-up times, multivariate regression analysis is performed. All calculations will be performed using SAS software.

ELIGIBILITY:
Inclusion criteria:

* A diagnosis of Epiretinal membrane,
* visual complaints consistent with Epiretinal membrane,
* age more than 50 years,
* refraction less than ± 5 diopters and astigmatism less than 3 diopters,
* indication for vitrectomy is only Epiretinal membrane.

Exclusion criteria:

* Previous intraocular surgery or laser-refractive procedure.
* Use of intraocular gas tamponade during the vitrectomy.
* Intraoperative manipulation of the intraocular lens.
* Serious complications (endophthalmitis, vitreous haemorrhage or retinal detachment).
* History of previous head or ocular trauma.
* Sulcus fixation of intraocular lens

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Refractive Error | One year
  Prediction error of intraocular lens calculation (measured in diopters)
Corneal endothelial count | One year
  measured in number of cells per square millimeter (mm2)
Macula anatomy | One year
  Macula-anatomy success of surgery, i.e. the postoperative decrease of macula thickness or postoperative macular oedema. Measured in millimeter.

SECONDARY OUTCOMES:
Anterior Chamber Depth | One year
  measured in millimeter (mm)
Axial length | One year
  measured in millimeter (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Hamoudi, MD, Principal Investigator — Eye Department Glostrup Hospital
Locations (1):
- Eye Department Glostrup Hospital, Glostrup Municipality, DK, Denmark